CLINICAL TRIAL: NCT04239248
Title: "Tasty&Healthy" is Not a Diet But a Dietary Approach: Randomized Controlled Trials of Excluding Pro-inflammatory Nutrients for Inducing and Maintaining Remission in Crohn's Disease
Brief Title: "Tasty&Healthy" Dietary Approach for Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tasty&Healthy
Record Dates: First submitted 2019-11-27; First posted 2020-01-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ACTIVE-RCT-I Tasty&Healthy intervention group (Experimental): Patients with mild-moderately symptomatic disease, will follow the Tasty&Healthy dietary approach.
  Interventions: Dietary Supplement: Tasty&Healthy intervention group
- ACTIVE-RCT-I Control group (Active Comparator): Patients with mild-moderately symptomatic disease, will receive EEN with Modulen formula only.
  Interventions: Dietary Supplement: EEN intervention group
- MH-RCT-II Tasty&Healthy intervention group (Experimental): Patients with laboratory evidence of mucosal inflammation but who are asymptomatic or have only minimal symptoms not requiring immediate treatment modification, will follow the Tasty&Healthy dietary approach.
  Interventions: Dietary Supplement: Tasty&Healthy intervention group
- MH-RCT-II Control group (No Intervention): Patients with laboratory evidence of mucosal inflammation but who are asymptomatic or have only minimal symptoms not requiring immediate treatment modification, will continue their habitual diet.

INTERVENTIONS:
Dietary Supplement: Tasty&Healthy intervention group — patients will receive dietary advice to exclude pro-inflammatory dietary components based on the book "Tasty&Healthy".
  Arms: ACTIVE-RCT-I Tasty&Healthy intervention group; MH-RCT-II Tasty&Healthy intervention group
Dietary Supplement: EEN intervention group — Oral exclusive feeding of formulated food (EEN), using Modulen formula only, for 8 weeks in amount based on the Daily Recommendations Intake. Those not tolerating oral EEN can receive EEN via a nasogastric tube.
  Arms: ACTIVE-RCT-I Control group

SUMMARY:
Despite the advent of multiple novel medications, many patients with Crohn's disease (CD) fail to achieve mucosal healing (MH). Exclusive enteral nutrition (EEN) has been shown to induce clinical remission accompanied by MH in many of CD patients. The aim of this proposal is to explore the effectiveness of the "Tasty&Healthy" dietary approach based on avoiding "pro-inflammatory" and processed ingredients, for inducing and maintaining remission and MH in children and young adults. This approach is based on the previously published charity cook-book "Tasty&Healthy" and might be more feasible than currently available nutritional treatments in CD. It does not offer a rigid diet with specific nutrients and does not require concurrent use of a formula feed.

The investigators hypothesize that a flexible dietary intervention of excluding processed and pro-inflammatory ingredients will improve the rate of clinical remission and MH without the need for liquid formula or structured rigid diet which are more difficult to adhere to. The investigators also hypothesize that home kits of Fecal calprotectin (FC), can personalize the diet thereby increasing feasibility for maintenance therapy in some patients.

DETAILED DESCRIPTION:
The investigators plan to conduct a set of three studies: Two randomized controlled trials (RCT) both including the Tasty&Healthy dietary intervention for 8 weeks in CD patients aged 6-24 years vs. 1) EEN in mild-moderate CD, and the other RCT in CD patients aged 6-40 years vs. 2) a control group continuing their habitual diet in those with mucosal inflammation despite stable medical treatment, but who are in clinical remission or have only minimal symptoms not requiring immediate treatment.

As a third study, responders from both trials will be offered to participate in an open label extension personalized-diet study of further 16 weeks (total 24 weeks), in which gluten and dairy will be gradually re-introduced based on repeated monthly home assays of FC while otherwise following the Tasty&Healthy dietary intervention in a treat-to-target management approach.

Patients will be evaluated at baseline, week 4 and week 8 with additional weekly phone visits to ensure adherence with the diets and address questions.

The extension study will include two clinic visits at weeks 16 and 24 and a monthly call to ensure adherence.

The investigators hope to establish a dietary-approach which is simpler to implement than current nutritional alternatives. It will enable high flexibility in the allowed foods and does not require liquid formula. In turn, this could position Tasty&Healthy, not merely for inducing remission, but also as a feasible maintenance strategy in selected patients.

ELIGIBILITY:
Inclusion Criteria:

ACTIVE-RCT-I

1. Children and young adults aged 6-24 years with established diagnosis of CD by European crohn's and colitis organisation (ECCO) /The European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) criteria.
2. <1 years of disease duration since the time of CD diagnosis.
3. Willingness to provide stool samples during the visits, at baseline, week 4 and week 8.
4. Mild- moderate disease activity (wPCDAI 20-57.5 or CDAI 200-45) or milder disease (wPCDAI 12.5-57.5 or CDAI 150-450) that according to the physician's discretion warrants an immediate change in treatment (and thus cannot be included in the MH-RCT-II that has a non-treatment arm).
5. Currently receiving no drug treatment or on maintenance treatment with immunomodulators (at stable dose for at least 16 weeks) or 5-aminosalicylic acid (5ASA)/sulfasalazine (at stable dose for at least 8 weeks). No current or prior treatment with biologics is allowed (i.e. biologic-naïve).

MH-RCT-II

1. Children and young adults aged 6-40 years with established diagnosis of CD by ECCO/ESPGHAN criteria.
2. <1 years of disease duration since the time of CD diagnosis, or <3 years of disease duration since the time of CD diagnosis for patients without evidence of significant bowel wall thickening (≤4 mm) without any damage as much as known.
3. Willingness to provide stool samples during the visits, at baseline, week 4 and week 8.
4. MINI ≥8 points.
5. Clinical remission or at most minimal symptoms (wPCDAI<20/ CDAI<200) that according to the physician's discretion do not warrant immediate medical treatment.
6. Receiving no treatment or on maintenance treatment with immunomodulators and/or first biologic (both at stable dose and interval for at least 16 weeks), and/or 5ASA/sulfasalazine (at stable dose for at least 8 weeks).

Second line biologics are allowed for patients without evidence of significant bowel wall thickening (≤4 mm) without bowel damage as much as known.

Exclusion Criteria:

1. Fibrostenotic or penetrating phenotype.
2. Fistulizing perianal disease which is not in complete remission.
3. "Ulcerative colitis (UC)-like" isolated Crohn's colitis.
4. Prior failure of exclusive enteral nutrition or any other dietary intervention, for any reason.
5. The use of steroids or budesonide in the recent month, or antibiotics prescribed to treat the CD in the previous two weeks.
6. Any formula feed during the last month.
7. Prior intestinal resection.
8. Pregnancy.
9. Celiac disease.
10. For ACTIVE-RCT-I: any prior or concurrent biologic therapy; for MH-RCT-II: any prior or concurrent biologic therapy other than second line biologic

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 129 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
ACTIVE-RCT-I: patient's tolerance to the diet by week 8. | 8 weeks
  Percent of patients tolerating the diet. Tolerance is defined as the absence of all of the three following items:
  1. Intolerance: cessation of dietary therapy because of patient's refusal to continue diet (based on reporting and the 24 hour recall);
  2. Poor adherence based on the modified Medication Adherence Report Scale (MARS) questionnaire; The modified MARS questionnaire rates How closely patients adhere to the diet. This is a self-report measure of adherence. It can be used to determine patients' willingness and ability to comply with the diet daily. A score of 1-5 indicates that the patient is not adherent; a score of 6-9 indicates that the patient is adherent.
  3. Poor adherence based on direct questioning (any answer other than "adheres to diet very often/always" will be considered poor compliant).
MH-RCT-II: Rate of mucosal healing (MH). | 8 weeks
  Percent of patients achieving MH defined by the proportion of patients with FC response as defined by reduction of at least 50% of FC levels from baseline; this has been added to the initial primary endpoint (i.e. MINI<8 points) after enrolling five patients given new data that the MINI is less accurate in adults.

SECONDARY OUTCOMES:
Percent of patients achieving MH rate at Week 8 assessed with panenteric capsule endoscopy (i.e. Crohn's capsule) at the end of both trials as the major secondary outcome. | 8 weeks
  Rate of MH defined by a central reading panel which will include leading irritable bowel disease (IBD) medical experts. This panel will determine the mucosal inflammation rate at week 8.
Percent of patients achieving clinical remission rate | 8 weeks
  Weighted Pediatric Crohn's Disease Activity Index (wPCDAI) by<12.5 points or Crohn's Disease Activity Index (CDAI)<150
Response rate defined as percent of patients achieving clinical remission and either reduction of FC levels. | 8 weeks
  Clinical remission: wPCDAI by<12.5 points or CDAI<150, and either reduction of at least 50% of FC levels from baseline or FC levels<150 µgr/gr.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Aharoni-Frutkoff Y, Plotkin L, Pollak D, Livovsky J, Focht G, Lev-Tzion R, Ledder O, Assa A, Yogev D, Orlanski-Meyer E, Broide E, Kierkus J, Kang B, Weiss B, Aloi M, Schwerd T, Shouval DS, Bramuzzo M, Griffiths AM, Yassour M, Turner D. Whole Food Diet Induces Remission in Children and Young Adults With Mild to Moderate Crohn's Disease and Is More Tolerable Than Exclusive Enteral Nutrition: A Randomized Controlled Trial. Gastroenterology. 2025 Dec;169(7):1462-1474.e2. doi: 10.1053/j.gastro.2025.06.011. Epub 2025 Jun 17. PMID 40553742